CLINICAL TRIAL: NCT01824589
Title: Effects of Intrathoracic Pressure Regulation Therapy in Patients With Elevated Intracranial Pressure Due to Brain Injury or Intracranial Pathology
Brief Title: Effect of Intrathoracic Pressure Regulation on Traumatic Brain Injury
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Advanced Circulatory Systems (Industry)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ACSI W81XWH-11-1-0542; W81XWH-11-1-0542 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2013-03-29; First posted 2013-04-05 (Estimated); Results first posted 2015-02-16 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Head Injury
Keywords: traumatic brain injury; TBI; ITPR; intrathoracic pressure regulator; hepatic encephalopathy; pseudotumorcerebri; obstructive hydrocephalus; intracranial hemorrhage
MeSH Terms: conditions — Craniocerebral Trauma; Brain Injuries, Traumatic; Hepatic Encephalopathy; Hydrocephalus; Intracranial Hemorrhages

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A (Active Comparator): tidal volume setting of 6ml/kg with the -7cm H2O ITPR as first device
  Interventions: Device: -7 cm H2O ITPR
- Group B (Active Comparator): tidal volume setting of 8ml/kg with the -7cm H2O ITPR as first device
  Interventions: Device: -7 cm H2O ITPR
- Group C (Active Comparator): tidal volume setting of 6ml/kg with the -12cm H2O ITPR as first device
  Interventions: Device: -12cm H2O ITPR
- Group D (Active Comparator): tidal volume setting of 8ml/kg with the -12cm H2O ITPR as first device
  Interventions: Device: -12cm H2O ITPR

INTERVENTIONS:
Device: -7 cm H2O ITPR — Single use disposable non-invasive device that is connected to a vacuum source and a means to deliver a positive pressure breath and generates negative3 pressure during the expiratory phase, thus creating subatmospheric intrathoracic pressure of -7 cmH2O between periods of positive pressure ventilations.
  Other Names: Intrathoracic Pressure Regulator, CirQlator
  Arms: Group A; Group B
Device: -12cm H2O ITPR — Single use disposable non-invasive device that is connected to a vacuum source and a means to deliver a positive pressure breath and generates negative3 pressure during the expiratory phase, thus creating subatmospheric intrathoracic pressure of -12 cmH2O between periods of positive pressure ventilations.
  Other Names: Intrathoracic Pressure Regulatory, CirQlator
  Arms: Group C; Group D

SUMMARY:
The purpose of this study is to demonstrate proof of clinical concept that application of the Intrathoracic Pressure Regulator (ITPR) will result in an increase in Cerebral Perfusion Pressure (CPP) and a decrease in Intracranial Perfusion Pressure (ICP) in patients with head injury and elevated ICP, and to determine the optimal ventilation tidal volume (TV).

ELIGIBILITY:
Inclusion Criteria:

* ≥15 years of age
* intubated and mechanically ventilated on a volume controlled mode
* head injury or other intracranial pathology with ICP of ≥15 mmHg
* arterial line in place
* SpO2 ≥95%
* MAP >60
* in ICU or about to undergo neurosurgery with planned placement of an ICP monitor
* inclusion presents no significant delays to planned emergent neurosurgery
* prior written informed consent

Exclusion Criteria:

* cardiac or pulmonary injury impacting intrathoracic pressure
* confirmed pneumothorax or hemothorax
* PaO2/FiO2 <300
* serious neck injury resulting in neck swelling with jugular venous compression
* evidence of ongoing uncontrolled bleeding
* respiratory disease such as COPD, interstitial lung disease, or other parenchymal or pulmonary vascular disease
* congestive heart failure

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-08; Primary Completion 2012-08 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: no device (washout) with tidal volume setting of 6ml/kg for 20 minutes, then 6ml/kg with the -7cm H2O ITPR as first device for 15 minutes, then tidal volume increased to 8ml/kg with the -7cm H2O ITPR for 15 minutes, then no device with 8ml/kg for 20 minutes, then 8ml/kg with -12cm H2O ITPR for 15 minutes, then 6ml/kg with -12cm H2O ITPR for 15 minutes, then no device with 6ml/kg.
  -7 cm H2O ITPR: Single use disposable non-invasive device that is connected to a vacuum source and a means to deliver a positive pressure breath and generates negative3 pressure during the expiratory phase, thus creating subatmospheric intrathoracic pressure of -7 cmH2O between periods of positive pressure ventilations.
- Group B: no device (washout) with tidal volume setting of 8ml/kg for 20 minutes, then 8ml/kg with the -7cm H2O ITPR as first device for 15 minutes, then tidal volume decreased to 6ml/kg with the -7cm H2O ITPR for 15 minutes, then no device with 6ml/kg for 20 minutes, then 6ml/kg with -12cm H2O ITPR for 15 minutes, then 8ml/kg with -12cm H2O ITPR for 15 minutes, then no device with 8ml/kg.
  -7 cm H2O ITPR: Single use disposable non-invasive device that is connected to a vacuum source and a means to deliver a positive pressure breath and generates negative3 pressure during the expiratory phase, thus creating subatmospheric intrathoracic pressure of -7 cmH2O between periods of positive pressure ventilations.
- Group C: no device (washout) with tidal volume setting of 6ml/kg for 20 minutes, then 6ml/kg with the -12cm H2O ITPR as first device for 15 minutes, then tidal volume increased to 8ml/kg with the -12cm H2O ITPR for 15 minutes, then no device with 8ml/kg for 20 minutes, then 8ml/kg with -7cm H2O ITPR for 15 minutes, then 6ml/kg with -7cm H2O ITPR for 15 minutes, then no device with 6ml/kg.
  -12cm H2O ITPR: Single use disposable non-invasive device that is connected to a vacuum source and a means to deliver a positive pressure breath and generates negative3 pressure during the expiratory phase, thus creating subatmospheric intrathoracic pressure of -12 cmH2O between periods of positive pressure ventilations.
- Group D: no device (washout) with tidal volume setting of 8ml/kg for 20 minutes, then 8ml/kg with the -12cm H2O ITPR as first device for 15 minutes, then tidal volume decreased to 6ml/kg with the -12cm H2O ITPR for 15 minutes, then no device with 6ml/kg for 20 minutes, then 6ml/kg with -7cm H2O ITPR for 15 minutes, then 8ml/kg with -7cm H2O ITPR for 15 minutes, then no device with 8ml/kg.
  -12cm H2O ITPR: Single use disposable non-invasive device that is connected to a vacuum source and a means to deliver a positive pressure breath and generates negative3 pressure during the expiratory phase, thus creating subatmospheric intrathoracic pressure of -12 cmH2O between periods of positive pressure ventilations.
Period: Overall Study
Arm/Group | Group A | Group B | Group C | Group D
Started | 1 | 0 | 0 | 0
Completed | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group D | Total
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
Age, Categorical [Number; unit: participants]
  <=18 years | 0 |  |  |  | 0
  Between 18 and 65 years | 0 |  |  |  | 0
  >=65 years | 1 |  |  |  | 1
Gender [Number; unit: participants]
  Female | 0 |  |  |  | 0
  Male | 1 |  |  |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Intracranial Pressure (ICP)
Description: Change in ICP from baseline will be compared with the ICP during 15 minutes of ITPR use.
Time Frame: 15 minutes after device is activated
Measure: Number; unit: mmHg
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 1 | 0 | 0 | 0
mmHg
  6ml/kg; -7cmH2O | -1 |  |  |
  8ml/kg; -7cmH2O | -1 |  |  |
  8ml/kg; -12cmH2O | 4 |  |  |
  6ml/kg; -12cmH2O | NA — Protocol discontinued after 8ml/kg with -12cmH2O device as patient was not tolerating device |  |  |

2. Secondary Outcome: Cerebral Perfusion Pressure (CPP)
Description: Measurement of the difference between baseline CPP and CPP at 15 minutes
Time Frame: 15 minutes after device activation
Measure: Number; unit: mmHg
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 1 | 0 | 0 | 0
mmHg
  6ml/kg; -7cmH2O | -1 |  |  |
  8ml/kg; -7cmH2O | 1 |  |  |
  8ml/kg; -12cmH2O | -5 |  |  |
  6ml/kg; -12cmH2O | NA — Protocol discontinued after 8ml/kg with -12cmH2O due to patient not tolerating device |  |  |

3. Secondary Outcome: Lung Compliance
Description: Change in lung compliance following each ITPR treatment compared to baseline.
Time Frame: baseline and immediately after device removal
Measure: Number; unit: ml/cmH2O
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 1 | 0 | 0 | 0
ml/cmH2O
  6ml/kg; -7cmH2O | 5.6 |  |  |
  8ml/kg; -7cmH2O | 3.3 |  |  |
  8ml/kg; -12cmH2O | -0.7 |  |  |
  6ml/kg; -12cmH2O | NA — Protocol discontinued after 8ml/kg with -12cmH2O device as patient was no longer able to tolerate device |  |  |

4. Secondary Outcome: Arterial Blood Gases (PaCO2)
Description: Arterial blood gases will be collected.
Time Frame: 15 minutes after device activation
Measure: Number; unit: mmHg
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 1 | 0 | 0 | 0
mmHg
  6ml/kg; -7cmH2O | 45.0 |  |  |
  8ml/kg; -7cmH2O | 44.7 |  |  |
  8ml/kg; -12cmH2O | 44.4 |  |  |
  6ml/kg; -12cmH2O | NA — Protocol discontinued after 8ml/kg with -12cmH2O device as patient was no longer able to tolerate device |  |  |

ADVERSE EVENTS:
Arm/Group | Group A | Group B | Group C | Group D
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No